CLINICAL TRIAL: NCT02078011
Title: Treatment of Breast Fibroadenoma With High Intensity Focused Ultrasound (HIFU): A Feasibility Study
Brief Title: Treatment of Breast Fibroadenoma With High Intensity Focused Ultrasound
Acronym: HIFU-FA-001
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: David R. Brenin, MD (Other)
Collaborators: Theraclion SAS, Paris, France (Unknown)
Responsible Party: Sponsor-Investigator, David R. Brenin, MD, Associate Professor, Department of Surgery, University of Virginia
Organization: University of Virginia (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17277
Record Dates: First submitted 2014-02-25; First posted 2014-03-04 (Estimated); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Breast Fibroadenoma
MeSH Terms: conditions — Fibroadenoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HIFU treatment (Experimental): The high intensity focused ultrasound (HIFU) will be administered to the targeted site to create heat and cause the cells to die
  Interventions: Device: High Intensity Focused Ultrasound

INTERVENTIONS:
Device: High Intensity Focused Ultrasound — The Echopulse device is a computer driven system which uses ultrasound to guide a high intensity focused ultrasound beam to a targeted area (the fibroadenoma in the breast).
  Other Names: Echopulse

SUMMARY:
The purpose of this study is to test an investigational device called the Echopulse for treatment of breast fibroadenomas in women. Fibroadenomas are benign (noncancerous) breast tumors that are made of glandular and fibrous breast tissue. These lumps can occur alone, in groups, or as a complex of lumps together. Sometimes women feel these in the breast when doing regular self breast exams, or they may be found during a routine mammogram. Some are small (less than an inch in size), and others are quite large (the size of a lemon or larger).

This is a study about the Echopulse device, a computer driven system which uses ultrasound to guide a high intensity focused ultrasound beam to a targeted area (the fibroadenoma in the breast). The high intensity focused ultrasound (HIFU) heats the targeted site which causes the cells to die and allows the possibility to treat the fibroadenoma without the need for surgery.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of fibroadenoma with histological confirmation of fibroadenoma of the breast
* Fibroadenoma is palpable
* Fibroadenoma is 1 cm or greater at its largest dimension and no less than 9 mm in the anterior-posterior dimension
* Fibroadenoma volume is between 2 cc and 10 cc
* Patient must give written informed consent (personally signed and dated) before completing any study-related procedure

Exclusion Criteria:

* Patient is pregnant or nursing
* Patient with breast implants in the target breast
* Patient with a breast cyst within the fibroadenoma to be treated
* Patient participating in another clinical trial involving an investigational drug, device or biologic

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-04; Primary Completion 2016-08-29 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
Change in volume of fibroadenoma | baseline, 3, 6, and 12 months
  Fibroadenoma volume with be measured by ultrasound.
Size of fibroadenoma | baseline, 3, 6, and 12 months
  Fibroadenoma will be assessed by physical examination including measurement of tumor size at clinic visits.
Patient reported outcomes | up to 12 months
  Patient-rated pain and patient responses to Satisfaction Questionnaire will be measured at intervals up to 12 months following HIFU treatment session

SECONDARY OUTCOMES:
Incidence of adverse events | up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: David Brenin, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States